CLINICAL TRIAL: NCT03001102
Title: Preoperative Bath in Patients Submitted to Hip Arthroplasty: Randomized Clinical Trial
Brief Title: Preoperative Bath in Patients Submitted to Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Lucia Maciel de Castro Franco, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EE-UFMG
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Surgical Wound Infection
Keywords: Preoperative Care; Baths; Chlorhexidine; Soaps; Povidone-Iodine; Arthroplasty, Replacement, Hip; Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Abortion, Induced

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bathing with 4% Chlorhexidine gluconate (Sham Comparator): Two baths with chlorhexidine using precise methods, including to scrubb the whole body with 50mL of undiluted solution, at night before surgery and the morning of surgery.
  Interventions: Device: 4% Chlorhexidine gluconate
- Bathing with10% PVPI degermante (Experimental): Two baths with PVPI using precise methods, including to scrubb the whole body with 50mL of undiluted solution for each bath, at night before surgery and the morning of surgery.
  Interventions: Device: 10% PVPI degermante
- Bathing with soap without antiseptic. (Active Comparator): Two baths with soap using precise methods, including to scrubb the whole body with 50mL of undiluted solution for each bath, at night before surgery and the morning of surgery.
  Interventions: Device: Soap without antiseptic

INTERVENTIONS:
Device: 4% Chlorhexidine gluconate — Cationic biguanide - antimicrobial action rubbing in the skin.
  Other Names: HiBiScrub; 4% Chlorhexidine degermante
  Arms: Bathing with 4% Chlorhexidine gluconate
Device: 10% PVPI degermante — Polymer soluble in water of iodine with polyvinylpyrrolidone (PVP) - antimicrobial action rubbing in the skin.
  Other Names: Betadine; 10% Povidone iodine degermante
  Arms: Bathing with10% PVPI degermante
Device: Soap without antiseptic — Liquid soap with glycerin, neutral pH. Skin cleansing
  Other Names: Non-medicated soap; Soap
  Arms: Bathing with soap without antiseptic.

SUMMARY:
Clinical trial for prevention, randomized, controlled, blinded, parallel, with three arms which purpose is verify the effects of nursing intervention preoperative bathing with 4% chlorhexidine gluconate, 10% Povidone iodine (PVPI) and soap without antiseptic, for the prevention of surgical site infection (SSI) in patients undergoing hip arthroplasty.

DETAILED DESCRIPTION:
Despite the recommendation in several guidelines of preoperative bathing with 4% chlorhexidine gluconate as a measure for the prevention of SSI, there is no evidence in the literature that support this practice. The objective of this study is to evaluate the effect of nursing intervention: preoperative bath using 4% chlorhexidine gluconate solutions, 10% povidone iodine degermante or soap without antiseptic for the prevention of SSI in patients undergoing elective hip arthroplasty surgery. The specific objectives are to compare the incidence of SSI in the three interventions, to assess the most effective intervention for the prevention of surgical infection and to estimate the frequency of allergic reactions caused by the use of the solutions. Two intervention groups (4% Chlorhexidine gluconate and PVPI10%) and a control group (without antiseptic soap) composed of 52 patients undergoing hip arthroplasty in each group will be randomized to perform the baths in the period from may 2015 to june 2017. Before the intervention, nasal swabs will be collected of patients to investigate colonization by Staphylococcus aureus.

The expected result is lower ISC rate with the proposed measures.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 or older;
* Elective procedure of total hip arthroplasty
* No report of infectious focus at the surgical site
* Know to respond to the clinical signs of a surgical infection or having a person responsible with this ability
* Do not be a nasal carrier of Staphylococcus aureus before surgery
* Have access to fixed or mobile phone

Exclusion Criteria:

* Patient treating surgical site infection
* Emergency hip prosthesis surgery or orthopedic trauma
* Nasal carriers of Staphylococcus aureus before surgery
* Previous history of allergic reactions to the products used in the bat

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Infection of Surgical Site (SSI) | During the first 90 days after surgery
  The infections that develop after the surgical procedure

SECONDARY OUTCOMES:
Allergic reactions | In the first hours after procedure
  Adverse reaction to a given product

CONTACTS AND LOCATIONS:
Overall Officials: Lúcia MC Franco, PhD student, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
The study and the information provided will be confidential and used only for purposes of this research. Disclosure of information will be anonymous and in conjunction with the responses of a group of people, never individually.